CLINICAL TRIAL: NCT00934908
Title: Prevention of Weight Gain and Dyslipidemia by Green Tea in Patients Initiating Therapy With Olanzapine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Green Tea and Olanzapine
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2009-07

CONDITIONS: Bipolar Disorder; Schizophrenia
Keywords: Zyprexa®; Green Tea; ALL
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Non-active "sugar pill"
  Interventions: Other: Placebo
- 2 (Active Comparator): Green Tea Capsules
  Interventions: Dietary Supplement: Green Tea

INTERVENTIONS:
Dietary Supplement: Green Tea — Green tea capsules taken twice a day.
  Arms: 2
Other: Placebo — Non-active "sugar pill".
  Arms: 1

SUMMARY:
The purpose of this study is to determine if taking green tea capsules can help prevent weight gain in patients that start therapy with Zyprexa® (olanzapine).

DETAILED DESCRIPTION:
Atypical antipsychotic (AA) medications are associated with obesity, diabetes mellitus, dyslipidemia, and cardiovascular disease.1 The prevalence of obesity in the AA medicated population ranges from 40-60%, compared to 30% of the general population. Treatments that are aimed at either reducing the burden of obesity in psychotic illness or preventing the weight gain and other metabolic changes associated with AA are needed. One potential therapy that has received inadequate clinical evaluation is Green tea (Camillia sinensis; GT). GT contains flavonoids including epigallocatechin gallate (EGCG), as well as caffeine, that have been documented to promote weight and fat loss in normal to overweight healthy subjects. Recently green tea was shown to significantly decrease plasma LDL and triglyceride concentrations and increase HDL concentrations in obese women. GT has never been evaluated for its potential to prevent weight gain or changes in plasma lipid concentrations in patients initiating therapy with AA. However, case reports of individuals indicate that treatment with a green tea extract may have efficacy in preventing weight gain in 4 patients that initiated treatment with quetiapine.

We hypothesize that intake of GT in the form of a dietary supplement will result in significantly less weight gain than supplementation with placebo in patients initiating therapy with Zyprexa®. We propose to conduct an 12-week double-blind, placebo-controlled pilot study of 48 out-patient volunteers to determine if twice daily supplementation with GT 1) attenuates weight and fat gain in patients initiating therapy with Zyprexa® and 2) attenuates changes in cardiovascular risk factors including plasma lipoprotein and triglyceride concentrations. The experiments will be performed on patients who initiate therapy with Zyprexa® with a BMI < 40kg/m2 that do not have dyslipidemia requiring pharmacologic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Concurrently taking Zyprexa® for a psychiatric indication such as bipolar disorder or schizophrenia
* Stable body weight (+ 5%) for at least 2 weeks prior to baseline visit
* No weight loss program participation within past 3 months

Exclusion Criteria:

* Treatment with an atypical Anti-psychotic treatment other than olanzapine with the past 6 months
* BMI > 40 kg/m2
* Use of any dietary supplements related to weight gain or weight loss within past 1 month
* Use of any medication related to weight or plasma lipid concentration (other than hormonal contraceptives). This includes, but not limited to: antihypertensives, benzodiazepines statins, and psychostimulants.
* Uncontrolled hypertension (SBP >140 or DBP > 90 mmHg)
* Use of a hypertensive medication
* Known active alcohol or substance abuse or consumption of > three alcoholic beverages/day.
* Active cardiovascular disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Attenuation of weight and fat gain in patients initiating therapy with Zyprexa® | Weeks 1, 6 and 12

SECONDARY OUTCOMES:
Attenuation of negative changes in the plasma lipid profile in patients initiating therapy with Zyprexa®. | Weeks 1, 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Donovan, PhD, Principal Investigator — Medical University of South Carolina; Thomas W Uhde, MD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States